CLINICAL TRIAL: NCT03414437
Title: Post-eRADicAte: A Long Term Follow up to eRADicAte (NCT 02097303), an Open Label Phase Two Study of RADium Ra 223 Dichloride With Concurrent Administration of Abiraterone Acetate Plus Prednisone in CRPC Subjects With Symptomatic Bone Metastasis.
Brief Title: Post-eRADicAte - A Long Term Follow up of Subjects That Completed the eRADicAte Study (NCT 02097303)
Acronym: Post-eRADicAte
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Carolina Research Professionals, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: CRP-PCA-01.1
Record Dates: First submitted 2017-12-19; First posted 2018-01-30 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer Metastatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a Long Term Follow Up study to eRADicAte, an open label study designed to examine the effects of Radium Ra 223 dichloride with concurrent administration of Abiraterone Acetate plus Prednisone Castrate-Resistant (Hormone-Refractory) Prostate Cancer subjects with symptomatic bone metastasis.

DETAILED DESCRIPTION:
This is a Long Term Follow Up study to eRADicAte, an open label study designed to examine the effects on concurrent administration of Radium Ra 223 dichloride and Abiraterone Acetate plus Prednisone in subjects with symptomatic castrate resistant prostate cancer and with bone metastases.

31 subjects completed all study visits in the eRADicAte study, and were thus evaluable. All 31 subjects will be asked to participate in this Long Term Follow Up study which will evaluate overall survival, subsequent additional prostate cancer therapies and medications, radiographic changes and SSE's (Symptomatic Skeletal Events), incidence of bone marrow failure, and diagnosis with secondary malignancies.

Living subjects will be evaluated at least 12 weeks after their last dose of Radium Ra 223 dichloride and at each subsequent clinic visit. Deceased subject's data will be obtained retrospectively, from 12 weeks after the eRADicAte End of Treatment visit and prospectively through the date of death. The total duration of the study is expected to be 48 months

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects are adults over the age of 18 with mCRPC that completed the eRADicAte study. The living study subject or legally authorized representative must be able to understand and sign the written informed consent form.

Exclusion Criteria:

* A living study subject or his legally authorized representative are not able to understand or willing to sign the written informed consent form.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The evaluable population includes 31 subjects that completed the eRADicAte study. This population will be used for the analysis of the primary efficacy endpoint.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the overall survival of subjects that completed the "eRADicAte" study. | From the end of "eRADicAte" study, subjects will be followed retroactively from the time they completed the study and proactively for up to 4 years
  Long term follow up
To investigate subsequent prostate cancer therapies and medications of subjects that completed the "eRADicAte" study. | From the end of "eRADicAte" study, subjects will be followed retroactively from the time they completed the study and proactively for up to 4 years
  Long term follow up
To investigate radiographic changes of subjects that completed the "eRADicAte" study. | From the end of "eRADicAte" study, subjects will be followed retroactively from the time they completed the study and proactively for up to 4 years
  Long term follow up
To investigate SSE's of subjects that completed the "eRADicAte" study | From the end of "eRADicAte" study, subjects will be followed retroactively from the time they completed the study and proactively for up to 4 years
  Long term follow up
To investigate the incidence of bone marrow failure of subjects that completed the "eRADicAte" study. | From the end of "eRADicAte" study, subjects will be followed retroactively from the time they completed the study and proactively for up to 4 years
  Long term follow up
To investigate the occurence of subsequent diagnosis with secondary malignancies of subjects that completed the "eRADicAte" study. | From the end of "eRADicAte" study, subjects will be followed retroactively from the time they completed the study and proactively for up to 4 years
  Long term follow up

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Chesapeake urology Research Associates, Towson, Maryland
  - Urology Cancer Center and GU Research Network, Omaha, Nebraska
  - Associated Medical Professionals, Syracuse, New York
  - Oregon Urology Institute, Springfield, Oregon
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: No
31 subjects will be enrolled. The sample size is based on the number of subjects that completed the "eRADicAte" study. No statistical assumptions are made.